CLINICAL TRIAL: NCT03005353
Title: Randomized Clinical Trial for Treatment of Candidal Vulvovaginitis Using Cumin Seed Extract Vaginal Suppositories.
Brief Title: Treatment of Candidal Vulvovaginitis Using Cumin Seed Extract Vaginal Suppositories.
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, Dr, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CSE
Record Dates: First submitted 2016-12-23; First posted 2016-12-29 (Estimated); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Infection, Fungal
MeSH Terms: conditions — Mycoses | interventions — Clotrimazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cumin seed extract (Experimental): Group A (study group) will receive Cumin seed extract vaginal suppositories once daily for 7 days.
  Interventions: Drug: Cumin seed extract
- clotrimazole (Active Comparator): Group B will receive conventional clotrimazole vaginal suppositories once daily for 7 days.
  Interventions: Drug: clotrimazole

INTERVENTIONS:
Drug: Cumin seed extract — patients will receive the drug in suppository form
  Arms: Cumin seed extract
Drug: clotrimazole — patients will receive the drug in suppository form
  Arms: clotrimazole

SUMMARY:
Fungal infections have increased over the last two decades, largely because of the increasing size of the population at risk, including patients who are immunocompromised, broad-spectrum antibiotics and intravascular catheter users. Essential oils and other extracts of plants have evoked interest as sources of natural products. They have been shown to possess antibacterial, antifungal, antiviral, insecticidal and antioxidant properties. To the best of our knowledge, no study has examined the efficacy of cumin seed extract on relieving vulvovaginal candidiasis in vivo.

ELIGIBILITY:
Inclusion Criteria:

1. Women were 18-49 years old and were married;
2. They had not used antibiotics, immunosuppressive drugs, or vaginal drugs 14 days before the study;
3. They did not suffer from trichomonal vaginitis, bacterial vaginitis, or cervicitis based on direct smear;
4. Candidiasis culture was in agreement with clinical symptoms and patient's complaints.

Exclusion Criteria:

1. Pregnant and lactating women;
2. Those who had abnormal uterine bleeding;
3. Women with diabetes or autoimmune diseases;
4. Women refuse to participate in the study.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
The percentage of patients with complete cure | one week
  cure is defines as absence of symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No